CLINICAL TRIAL: NCT02297191
Title: Ultrasound Guided Local Anesthetic Field Block Within the Thoracolumbar Interfascial Plane: Distribution of Pain and Temperature Sensation Loss in Healthy Volunteers
Brief Title: Ultrasound Guided Local Anesthetic Block: Thoracolumbar Interfascial Plane
Acronym: TLIP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TLIP Block; Pro00033609 (Other: Medical University of South Carolina)
Record Dates: First submitted 2014-07-28; First posted 2014-11-21 (Estimated); Last update posted 2018-06-20 (Actual); Status verified 2016-03

CONDITIONS: Healthy
Keywords: volunteer; pilot study; adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Thoracolumbar Interfascial Plane Block (Experimental): All participants will have two injections at the same vertebral level on each side of the back. Each injection will consist of four 5cc incremental injections with aspiration prior to each 5cc of injectate of 0.5% Ropivicaine. . Each side of the back will be injected with 20cc of .05% Ropivicaine. Ultrasound will be used in real time to guide the needle, evaluate for "spread" of local anesthesia and to minimize the risk of Ropivicaine being injected intravascularly.
  a. Ultrasound images will be saved using the nomenclature TLIP Anat
  Interventions: Procedure: Thoracolumbar Interfascial Plane Block; Drug: Ropivicaine

INTERVENTIONS:
Procedure: Thoracolumbar Interfascial Plane Block — All participants will have two injections at the same vertebral level on each side of the back. Each injection will consist of four 5cc incremental injections with aspiration prior to each 5cc of injectate of 0.5% Ropivicaine. . Each side of the back will be injected with 20cc of .05% Ropivicaine. Ultrasound will be used in real time to guide the needle.
  1. Ultrasound images will be saved using the nomenclature TLIP Anatomy
  2. Photos will only include surface anatomy of the low-to-mid back.
  3. Participants will be assessed for evidence of adverse reaction to local anesthesia (tinnitus, disorientation, or perioral numbness) with each 5cc dose of local anesthetic. If any adverse reactions are noted the dosing will be stopped.
Drug: Ropivicaine

SUMMARY:
The purpose of the study is to determine the effectiveness of a new approach to numbing (anesthetizing) nerves in the back and to measure how far the area of anesthesia extends on the skin of the back.

DETAILED DESCRIPTION:
This research aims to define a novel field-infiltration nerve block. We will use ultrasound guidance to inject local anesthesia into the potential space between the muscle bodies of the erector spinae. The medial branch of the dorsal ramus of each thoracolumbar nerve innervates the muscle and skin overlying the erector spinae muscle to the midline. By anesthetizing each nerve we believe minimally invasive (1-2 level) back surgery may be completed with less pain and preclude the side-effect laden opioid analgesics.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Adult

Exclusion Criteria:

* Pregnant women (a urine pregnancy test will be done on all females of childbearing age)
* Liver dysfunction
* Elderly
* Impaired cardiovascular function
* Individuals on amiodarone or history of back surgery
* History of medical allergy to local amide type local anesthetics
* Medical allergy to chlorhexidine
* History of paresthesias
* Inability to lay flat
* Home oxygen requirement
* History of seizures
* Only adults will be eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-07; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Anesthesia (monitoring of pain, temperature, and adverse reaction to anesthesia [tinnitus, disorientation, or perioral numbness]) | The day of procedure (up to 15 minutes)
  At time zero (pre injection), 5 minutes, and 15 minutes point-discrimination to pain and temperature will be evaluated by blunt-needle prick and ice (in plastic bag). A "map" of each will be drawn and photographed for analysis.
  1. Photos will only include surface anatomy of the low-to-mid back.
  2. Participants will be assessed for evidence of adverse reaction to local anesthesia (tinnitus, disorientation, or perioral numbness) with each 5cc dose of local anesthetic.

CONTACTS AND LOCATIONS:
Overall Officials: William Hand, MD, Principal Investigator — Medical University of South Carolina; Scott T Reeves, MD, Study Chair — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Derived] Hand WR, Taylor JM, Harvey NR, Epperson TI, Gunselman RJ, Bolin ED, Whiteley J. Thoracolumbar interfascial plane (TLIP) block: a pilot study in volunteers. Can J Anaesth. 2015 Nov;62(11):1196-200. doi: 10.1007/s12630-015-0431-y. Epub 2015 Jul 7. PMID 26149600